CLINICAL TRIAL: NCT05929495
Title: Phase 2, Open-label, Single-arm Study on the Use of Metformin as Adjunctive Therapy in High-grade Glioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBM MET
Record Dates: First submitted 2023-06-13; First posted 2023-07-03 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma, IDH-wildtype; Metformin; Malignancies
Keywords: Metformin; Gliomas; GBM
MeSH Terms: conditions — Glioblastoma; Neoplasms; Glioma | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Metformin dose of 1 g/day orally in two administrations (500 mg tablets) during the first two weeks of treatment, increasing to 2 g/day in two 1 g tablets thereafter
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin (Experimental): 25 patients with GBM will take 1g/day of Metformin (2 tablets of 500 mg) for two weeks and then take 2g/day of Metformin for a total of 6 weeks. At the end of 6 weeks, treatment with Metformin alone will be continued for 4 weeks.
  Thereafter, the second-phase Stupp protocol (adjuvant TMZ) + metformin is resumed continuously until the end of the enrollment period, i.e., 58 weeks from the start of treatment, for each patient.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — The investigator will identify potential participants and confirm the diagnosis of GBM. Subjects will be screened within 6 weeks before starting treatment.
  Treatment will involve:
  * Administration of the standard or partial Stupp protocol (Radiotherapy + Temozolomide) in combination with Metformin for 6 weeks,
  * Treatment with only Metformin for 4 weeks;
  * Resumption of adjuvant TMZ + Metformin treatment continuously until the end of the enrollment period.

SUMMARY:
About 75% of CNS malignant tumors are classified as gliomas and the IDH-wildtype glioblastoma (GBM) represents the most aggressive form among CNS malignancies.

This is a nationwide single-center phase II drug clinical trial with an approximate duration of 32 months.

The clinical trial will be single-arm to evaluate the biological activity and effects of metformin in combination with TMZ in patients with GBM.

DETAILED DESCRIPTION:
About 75% of CNS malignant tumors are classified as gliomas, tumors of neuroectodermal origin arising from glial cells or glial cell precursors. The World Health Organization classification distinguishes gliomas into low-grade gliomas (low-grade gliomas, grade I and II) and high-grade gliomas (high-grade gliomas, grade III and IV).

IDH-wildtype glioblastoma (GBM) represents the most aggressive form among CNS malignancies.

Over the past century, numerous epidemiological and experimental observations have reported a preventive and beneficial antitumor effect of metformin, which has suggested the possibility of using it as adjunctive therapy in many cancer subtypes, including GBM.

The aim of this study is to evaluate the effect of Metformin as adjuvant therapy to TMZ in the treatment of patients with GBM.

Patients will start with a Metformin dose of 1 g/day orally in two administrations (500 mg tablets) during the first two weeks of treatment, increasing to 2 g/day in two 1 g tablets thereafter.

The approximate total duration of the study is 32 months, and 25 patients will be enrolled

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed histologically confirmed GBM (WHO grade IV, IDH wild type) undergoing surgical resection;
* hypomethylation or hypermethylation of MGMT assessed post-surgery;
* adult patients (≥18 years), both sexes;
* Patients undergoing Stupp protocol including patients aged > 70 years performing the hypofractionated protocol and three weeks of chemotherapy;
* Karnofsky Performance Status (KPS)> 60 assessed post-surgery;
* life expectancy at least 6 months defined by size and location of lesion tumor;
* freely given written informed consent prior to any activity related to the study. Patients must be able to communicate with the investigator and comply with the study procedures;
* Women of childbearing age must test negative for pregnancy at enrollment and, if they have sexual intercourse, they must agree to use specific contraceptive methods. Female subjects of childbearing age, i.e., fertile, after menarche and until post-menopause unless they are permanently infertile, who are sexually active, must apply a highly effective method of birth control with a low failure rate (i.e., less than 1 percent per year), such as combined hormonal contraception (containing estrogen and progestin) combined with ovulation inhibition (oral intravaginal, or transdermal), progestin-only hormonal contraception associated with ovulation inhibition (oral, injectable, or implantable), intrauterine device (IUD), intrauterine hormone delivery system (IUS), bilateral tubal occlusion, vasectomized partner, or sexual abstinence, throughout the treatment period and for four weeks after the last dose of the study treatment. Hormonal methods other than levonorgestrel-containing devices or medroxyprogesterone injections should be supplemented with the use of a male condom. Women of nonfertile age may be included if surgically sterile or postmenopausal for at least 2 years. The investigator is responsible for determining whether the patient has adopted an appropriate method of contraception for participation in the study.
* Male subjects with female partners of childbearing age must use condoms during treatment and until the end of relevant systemic exposure.

Exclusion Criteria:

* Multicenter GBMs;
* Patients diagnosed with diabetes or diabetes-related conditions;
* other active malignancies;
* hypersensitivity, intolerance to metformin or excipients;
* Impaired renal function with creatinine clearance < 60 mL/min assessed at recruitment, liver failure assessed at recruitment by clinical history and examination of ALT, AST and total bilirubin, and other contraindications to metformin use;
* taking metformin, insulin or other biguanides, regardless of the reason;
* pregnancy or lactation;
* patient has serious pre-existing medical conditions that, in the opinion of the investigator, would preclude participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Value of PFS at 6 months after the start of treatment | Frome baseline to 6 months
  It allow us to determine the efficacy at the recommended dose (RD) of metformin in patients with GBM

SECONDARY OUTCOMES:
EORTC QLQ-C30 questionnaire at 6 months after the start of treatment | Frome baseline to 6 months
  The Quality of Life of Cancer Patients questionnaire allow us to evaluate the change in the level of health-related quality of life.
  It consists of several questions that the patient must answer by choosing a value from 1 (minimum) to 4/7 (maximum), depending on the question.
MMSE questionnaire at 6 months after the start of treatment | Frome baseline to 6 months
  The Mini Mental State Evaluation questionnaire allow us to evaluate the change in the level of health-related quality of life.
  It consists of several questions for the patient to answer, but there are no minimum or maximum values for the patient to choose from.
Safety and tolerability assessment of treatment | From baseline through study completion, an average of 32 months
  Safety will be assessed throughout the study as type, frequency and severity of grade III and IV events.
  Tolerability will be assessed as number of discontinuations or dose reduction and by evaluation of clinical and hematochemical parameters
Plasma measurement of circulating metabolites | At study completion, an average of 32 months
  Peri-operative plasma will be taken from each patient for hematochemical analysis, in order to research of prognostic biomarkers.
Plasma measurement of adiponectin | At study completion, an average of 32 months
  Peri-operative plasma will be taken from each patient for hematochemical analysis, in order to research of prognostic biomarkers.
Proteomic analysis | At study completion, an average of 32 months
  Peri-operative plasma will be taken from each patient for proteomic analysis, in order to research of prognostic biomarkers.
Correlations between in vivo clinical response and effect of association measured in vitro on cell lines obtained from the same patient undergoing surgery | At the end of recruitment, an average of 18 months
  In vitro cell response measured as cell growth inhibition and correlation with clinical response (PFS) of the same patient.
Gene expression analysis | At the end of recruitment, an average of 18 months
  Identifying the molecular phenotype of cells taken from patients' tissue samples during surgery and comparing clinical response and molecular phenotype by transcriptomic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No